CLINICAL TRIAL: NCT05567562
Title: Dual Anti-platelet Therapy in Chronic Obstructive Pulmonary Disease Study
Brief Title: Anti-Platelets in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Carrie Pistenmaa, M.D, Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 2022P002327; K23HL141651 (NIH)
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: COPD; Emphysema; Emphysema or COPD
Keywords: Platelet Dysfunction; Pulmonary Blood Vessel Injury; COPD; Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema | interventions — Dual Anti-Platelet Therapy; Aspirin; Clopidogrel

STUDY DESIGN:
Intervention Model Description: Double-blind crossover study is a Phase 2 interventional study to assess whether dual-anti platelet therapy improves pulmonary blood flow compared to placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants, investigators and care providers will be blinded as to dual-anti platelet therapy or placebo treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- COPD Cases: Dual antiplatelet therapy first, then placebo (Experimental): Dual antiplatelet therapy (aspirin 81mg and clopidogrel 75mg) will be given for 2 weeks, followed by 2 weeks without intervention, then 2 weeks of placebo
  Interventions: Combination Product: dual anti-platelet therapy; Drug: Placebo
- COPD Cases: Placebo first, then dual antiplatelet therapy (Placebo Comparator): Placebos for each therapy (2 pills) will be given for 2 weeks, followed by 2 weeks without intervention, then 2 weeks of dual antiplatelet therapy
  Interventions: Combination Product: dual anti-platelet therapy; Drug: Placebo
- Controls: Dual antiplatelet therapy first, then placebo (Active Comparator): Dual antiplatelet therapy (aspirin 81mg and clopidogrel 75mg) will be given for 2 weeks, followed by 2 weeks without intervention, then 2 weeks of placebo
  Interventions: Combination Product: dual anti-platelet therapy; Drug: Placebo
- Controls: Placebo first, then dual antiplatelet therapy (Placebo Comparator): Placebos for each therapy (2 pills) will be given for 2 weeks, followed by 2 weeks without intervention, then 2 weeks of dual antiplatelet therapy
  Interventions: Combination Product: dual anti-platelet therapy; Drug: Placebo

INTERVENTIONS:
Combination Product: dual anti-platelet therapy — dual anti-platelet therapy
  Other Names: aspirin 81mg EC tab; clopidogrel 75mg tab
Drug: Placebo — Placebo

SUMMARY:
This is a 6 week crossover study in current and former smokers with and without COPD to evaluate whether 2 weeks of dual antiplatelet therapy (aspirin 81mg and clopidogrel 75mg) improves pulmonary perfusion (i.e. blood flow in the lungs measured on a contrast CT scan) compared to placebo.

DETAILED DESCRIPTION:
This is a single-center Phase IIa randomized double-blind crossover study in smokers with and without chronic obstructive pulmonary disease (COPD) to test whether dual antiplatelet therapy (aspirin 81mg and clopidogrel 75mg) improves pulmonary perfusion (i.e. blood flow in the lungs) compared to placebo.

We will enroll 30 subjects (20 with COPD, 10 without) who will each take part for 6 weeks. Participants and researchers will be blinded, they will not know which medications they are on first. Each participant will be asked to take aspirin and clopidogrel together for 2 weeks and also matching placebos for 2 weeks, with a 2 week washout period in between. Pulmonary blood flow will be evaluated with a contrast-enhanced CT scan of the chest two times over the 6 week study.

ELIGIBILITY:
Inclusion Criteria - COPD Cases:

* COPD (FEV1/FVC < 0.7, FVC >= LLN), GOLD Stage I/II/III (FEV1 >= 40%)
* Current or former smoker of at least 10 pack years

Inclusion Criteria - Controls:

* Normal lung function (FEV1/FVC >= 0.7, FEV1 and FVC >= LLN)
* Current or former smoker of at least 10 pack years

Exclusion Criteria:

* Platelet count < 150,000/dL or self-report of a bleeding disorder;
* Regular use of aspirin, clopidogrel or another antiplatelet medication;
* Allergy to aspirin, clopidogrel, albuterol or iodine/IV contrast;
* BMI > 35;
* History of intracranial hemorrhage, severe GI bleed or other life-threatening bleed;
* Use of blood thinner (e.g. warfarin, lovenox or novel oral anti-coagulants);
* Continuous use of supplemental oxygen at home;
* Regular use of an NSAID;
* Daily use of oral steroids, theophylline, roflumilast, or loop diuretics;
* History of organ transplant or autoimmune disease on systemic therapy (rheumatoid arthritis, lupus);
* Use of a biologic medication with regular injections;
* Other current lung disease (interstitial lung disease, idiopathic pulmonary fibrosis, asthma);
* IV drug use within the last year;
* History of lung surgery to remove part of the lung;
* Known bullae or advanced destructive emphysema in more than 1/3 of the lungs;
* Treatment for cancer (systemic therapy or surgical/radiation within the thorax) in the last 12 months;
* Known diagnosis of pulmonary hypertension;
* Known systolic heart failure (RV or LV EF < 40%);
* Acute or chronic renal insufficiency (estimated glomerular filtration rate [GFR] <60 mL/min/1.73 m2 or self-report). GFR will be calculated using the CKD-EPI equation;
* Current or planned pregnancy in the next year;
* Regular marijuana smoking;
* Exacerbation of respiratory symptoms within the previous 6 weeks, such as that requiring hospitalization, oral prednisone or antibiotics to control symptoms, or longer and not yet returned to baseline; and
* Chest, abdominal or eye surgery, or a heart attack or stroke, within the last 3 months.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Pulmonary microvascular blood volume, CV | 6 weeks
  Coefficient of variation (CV) of pulmonary microvascular blood volume on dual energy CT scan, comparing on dual antiplatelet therapy to placebo

SECONDARY OUTCOMES:
Pulmonary microvascular blood volume | 6 weeks
  Pulmonary microvascular blood volume on dual energy CT scan, comparing on dual antiplatelet therapy to placebo
Oxygen saturation | 6 weeks
  Resting oxygen saturation

OTHER OUTCOMES:
Vascular pruning on CT | 6 weeks
  Distal macrovascular pruning on non-contrast inspiratory CT
Percent emphysema on CT | 6 weeks
  Percent emphysema-950 on non-contrast inspiratory CT
Functional small airways disease on CT | 6 weeks
  Functional small airways disease, calculated from gas trapping on non-contrast expiratory and inspiratory CT
Lung function | 6 weeks
  Spirometry measures of forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and FEV1/FVC
Platelet activation measures | 6 weeks
  Platelet activation measures by flow cytometry: circulating monocyte-platelet aggregates (unstimulated), activated GPIIb/IIIa receptor, unstimulated, and stimulated by low and high dose arachidonic acid and adenosine diphosphate, and P-selectin on the platelet surface, unstimulated, and stimulated by low and high dose arachidonic acid and adenosine diphosphate. Also urine 11d-TXB2, plasma TXB2 and aspirin-triggered lipoxin A4
FeNO | 6 weeks
  Fraction of exhaled nitric oxide

CONTACTS AND LOCATIONS:
Overall Officials: Carrie L Pistenmaa, MD, MS, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
This is a small single-center study, we do not plan to share participant level data